CLINICAL TRIAL: NCT04888390
Title: The Effect of Exercise Intervention on Cardiorespiratory Function and Exercise Capacity in Heart Failure Patients With Diabetes Mellitus.
Brief Title: Exercise Intervention on Cardiorespiratory Function in HF With DM.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Kun-Ling Tsai, Associate Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-BR-110-016
Record Dates: First submitted 2021-05-05; First posted 2021-05-17 (Actual); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Heart Failure
Keywords: Heart failure; Diabetes mellitus; Exercise intervention; Cardiac rehabilitation
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study population will be randomized and separated in two groups, Intervention and Usual care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive multi-model exercise intervention 2-3 times per week for 3 months.
  Interventions: Behavioral: Muti-model exercise intervention
- Usual care group (Active Comparator): The Usual care group will receive heart failure disease and exercise-related education.
  Interventions: Behavioral: Disease and exercise suggestion

INTERVENTIONS:
Behavioral: Muti-model exercise intervention — The Muti-model exercise intervention include aerobic exercise training by ergometer or treadmill, resistance exercise by using elastic band and flexibility exercise by active stretch. The total training program takes for 60 minutes, 2-3 times per week for 3 months.
  Arms: Intervention group
Behavioral: Disease and exercise suggestion — The participants will be provided by educational program about heart failure self-care and home-based exercise approach.
  Arms: Usual care group

SUMMARY:
Investigate the effects of exercise training on the cardiopulmonary function and exercise capacity in diabetes mellitus with heart failure.

DETAILED DESCRIPTION:
This research intends to explore the effects of exercise training on the cardiopulmonary function and exercise tolerance of heart failure patients with diabetes mellitus. In addition to the impaired cardiac function, the clinical manifestations of patients with heart failure also shown the inefficiency of pulmonary function, peripheral vascular function, and musculoskeletal system. Due to low exercise tolerance, functional activities and quality of life are impaired. With the high hospitalization rate and high mortality rate, the clinical treatment of heart failure is challenging. At present, exercise has been listed in the guidelines for the treatment of heart failure, and is recommended that patients with heart failure should take regular aerobic exercise training to maintain functional activity and reduce symptoms. Past studies have also suggested that exercise training can help reduce the risk factors of cardiovascular disease and improve part of the cardiovascular function. Furthermore, exercise can improve the quality of life and reduce the hospitalization rate. Although diabetes is a common comorbidity of heart failure, and is a poor prognostic factor that increases the overall risk of heart failure and cardiovascular death, there are few studies in the past to further explore the benefits of exercise training for diabetes with heart failure, although current studies have confirmed that regular exercise can effectively control diabetes. However, the cardiopulmonary function and exercise tolerance of exercise training for diabetes with heart failure still need to be clarified. Therefore, this study aims to investigated the effect of cardiopulmonary function and exercise tolerance in patients with heart failure. The study participants were divided into two groups: usual care group and exercise group. Exercise training involved last for twelve weeks, and then follow up until the sixth week after exercise training. The results of the study are expected to be applied to clinical heart failure rehabilitation. It is expected that through active cardiopulmonary rehabilitation combined with precise and personalized exercise prescriptions, it will prevent deterioration of heart failure and may help improve the clinical practice of heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Heart Failure (NYHA I-III) with diabetes mellitus
* Aged 30-85
* Mini-mental state examination score > 25

Exclusion Criteria:

* eGFR < 30mL/min/1.73m2
* Exercise intervention contraindication of heart failure
* Pregnancy
* Uncontrolled disease

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
NT-proBNP | Change from baseline (0 week) to mid-intervention (6 weeks)
  N-terminal pro-brain natriuretic peptide
NT-proBNP | Change from baseline (0 week) to post-intervention (12 weeks)
  N-terminal pro-brain natriuretic peptide
NT-proBNP | Change from baseline (0 week) to follow up (24 weeks)
  N-terminal pro-brain natriuretic peptide
Oxygen consumption (VO2) | Change from baseline (0 week) to mid-intervention (6 weeks)
  Oxygen consumption examined by cardiopulmonary exercise test
Oxygen consumption (VO2) | Change from baseline (0 week) to post-intervention (12 weeks)
  Oxygen consumption examined by cardiopulmonary exercise test
Oxygen consumption (VO2) | Change from baseline (0 week) to follow up (24 weeks)
  Oxygen consumption examined by cardiopulmonary exercise test

SECONDARY OUTCOMES:
Quality of life score (Minnesota Living With Heart Failure Questionnaire) | Change from baseline (0 week) to mid-intervention (6 weeks)
  Heart Failure Questionnaire
Quality of life score (Minnesota Living With Heart Failure Questionnaire) | Change from baseline (0 week) to post-intervention (12 weeks)
  Heart Failure Questionnaire
Quality of life score (Minnesota Living With Heart Failure Questionnaire) | Change from baseline (0 week) to follow up (24 weeks)
  Heart Failure Questionnaire
FEV1/FVC | Change from baseline (0 week) to mid-intervention (6 weeks)
  Pulmonary function test
FEV1/FVC | Change from baseline (0 week) to post-intervention (12 weeks)
  Pulmonary function test
FEV1/FVC | Change from baseline (0 week) to follow up (24 weeks)
  Pulmonary function test
MIP (maximal inspiratory pressure) | Change from baseline (0 week) to mid-intervention (6 weeks)
  Inspiratory muscle function assessed by pressure meter
MIP (maximal inspiratory pressure) | Change from baseline (0 week) to post-intervention (12 weeks)
  Inspiratory muscle function assessed by pressure meter
MIP (maximal inspiratory pressure) | Change from baseline (0 week) to follow up (24 weeks)
  Inspiratory muscle function assessed by pressure meter
MEP (maximal exspiratory pressure) | Change from baseline (0 week) to mid-intervention (6 weeks)
  Inspiratory muscle function assessed by pressure meter
MEP (maximal exspiratory pressure) | Change from baseline (0 week) to post-intervention (12 weeks)
  Inspiratory muscle function assessed by pressure meter
MEP (maximal exspiratory pressure) | Change from baseline (0 week) to follow up (24 weeks)
  Inspiratory muscle function assessed by pressure meter

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ling Tsai, Ph.D., Principal Investigator — Department of Physical Therapy, National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD sharing plan will be decided after summarized data being published.